CLINICAL TRIAL: NCT02573831
Title: The Effect of Oxycodone to the Placental Circulation at Early Labour
Acronym: oksisynnII
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Kuopio University Hospital (Other)
Collaborators: Admescope Ltd (Industry)
Responsible Party: Principal Investigator, Merja Kokki, MD, PhD, Kuopio University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KUH12012015
Record Dates: First submitted 2015-10-08; First posted 2015-10-12 (Estimated); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Labor Pain
Keywords: labor; pain; oxycodone; placenta
MeSH Terms: conditions — Labor Pain; Pain | interventions — Oxycodone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): The patients are given at first placebo and after one hour oxycodone 0,05 mg/kg if needed
  Interventions: Drug: Placebo
- Oxycodone (Experimental): The patients are given at first oxycodone 0,05 mg/kg and after one hour oxycodone 0,05 mg/kg if their pain in numerical rating scale from 0 to 10 is 5 or more
  Interventions: Drug: Oxycodone

INTERVENTIONS:
Drug: Oxycodone — The patients are given at first oxycodone 0,05 mg/kg and after one hour oxycodone 0,05 mg/kg if their pain in numerical rating scale from 0 to 10 is 5 or more
  Arms: Oxycodone
Drug: Placebo — The patients are given at first placebo and after one hour oxycodone 0,05 mg/kg if their pain in numerical rating scale from 0 to 10 is 5 or more
  Arms: Placebo

SUMMARY:
Oxycodone is used to treat pain in early labor, however the effect of oxycodone to placental or fetal circulation has not been evaluated. Oxycodone is increasingly used to treat labor pain in the early phase. The aim of the randomised, double blinded, placebo controlled study was to evaluate the effects of oxycodone in placental circulation, efficacy and safety of oxycodone and the effects to the newborn.

ELIGIBILITY:
Inclusion Criteria:

* oxycodone planned for pain relief

  * age 18 years or more
  * Informed consent obtained
  * Full term pregnancy

Exclusion Criteria:

* No oxycodone planned

  * age less than 18 years
  * No informed consent
  * not full term pregnancy
* Other contraindication to oxycodone

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2015-02-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
placental blood flow | from zero hours to two hours after the first study drug
  Placental blood flow is measured with doppler ultrasound

SECONDARY OUTCOMES:
uterine arterial flow | from zero hours to two hours after the first study drug
  uterine arterial flow is measured with doppler ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Merja Kokki, MD, PhD, Principal Investigator — Kuopio University Hospital
Locations (1):
- Kuopio University Hospital, Kuopio, Northern Savonia, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Alanne L, Kokki H, Mykkanen A, Orden MR, Rinne V, Rasanen J, Kokki M. Oxycodone does not affect placental circulatory physiology during the early first stage of labor-A randomized trial. Acta Obstet Gynecol Scand. 2023 Aug;102(8):1063-1072. doi: 10.1111/aogs.14603. Epub 2023 Jun 21. PMID 37344997